CLINICAL TRIAL: NCT06794008
Title: An Open, Single-Arm, Single-Center Clinical Study Assessing the Safety and Efficacy of BCMA-CD19 Targeted Chimeric Antigen Receptor T-Cell Therapy in Multiple Refractory Autoimmune Diseases
Brief Title: BCMA-CD19 CAR-T Therapy for Refractory Autoimmune Diseases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, He Jing, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICG318-AAV-02
Record Dates: First submitted 2025-01-06; First posted 2025-01-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-12

CONDITIONS: Systemic Lupus Erythematosus; Inflammatory Myopathy; Systemic Sclerosis (SSc); ANCA-associated Vasculitis; IgG4-Related Diseases; Antiphospholipid Syndrome; Acquired Thrombotic Thrombocytopenic Purpura; Behcet Disease; Sjogren Syndrome
Keywords: CAR-T; CD19; BCMA
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Myositis; Scleroderma, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Immunoglobulin G4-Related Disease; Antiphospholipid Syndrome; Purpura, Thrombotic Thrombocytopenic; Behcet Syndrome; Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T treatment in patients with multiple refractory autoimmune diseases (Experimental): Patients received the BCMA-CD19-targeted CAR-T cells with a dosage of 3×10^6/kg CAR-T cells per kilogram.
  Interventions: Drug: BCMA-CD19 CAR-T therapy

INTERVENTIONS:
Drug: BCMA-CD19 CAR-T therapy — Patients received the BCMA-CD19-targeted CAR-T cells with a dosage of 3×10^6/kg CAR-T cells per kilogram.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of BCMA/CD19 chimeric antigen receptor (CAR)-modified T cells in the treatment of autoimmune diseases.

DETAILED DESCRIPTION:
The investigators designed a single-center, open-label, single-arm clinical study. Adults with multiple refractory autoimmune diseases will be enrolled, meeting the inclusion criteria. BCMA-CD19 targeted chimeric antigen receptor T-cells will be administered intravenously 1-2 days after preconditioning, at a dose of 3×10^6/kg of CAR-T cells per kilogram (referring to successfully transduced CAR-T cells, not total T cells). The total volume of the CAR-T cell suspension administered per patient will range from approximately 10 to 70 mL, using a "single-dose" regimen. The entire dose of CAR-T cells will be infused intravenously rapidly on day 0. Patients will be evaluated for improvements in clinical and laboratory parameters to assess the safety and efficacy of BCMA-CD19 CAR-T therapy. The primary endpoints include the Complete Remission Rate and laboratory indicators. Secondary endpoints include pharmacokinetic characteristics, long-term efficacy, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age, 18-65 years old (inclusive), weight >=45kg, male and female;
2. The diagnosis of each disease meets the following criteria:

Systemic lupus erythematosus: 1997 ACR classification criteria or 2012 SLICC classification criteria Sjögren's syndrome: 2002 International Classification of Sjögren's Syndrome Inflammatory myopathies: 1977 Bohan Recommendation Systemic sclerosis: 1980 ACR classification criteria or 2013 ACR-EULAR classification criteria Behcet's disease: 1989 International Classification Criteria for Behcet's disease ANCA-associated vasculitis: 1990 ACR classification criteria IgG4-related disease: 2011 IgG4-RD composite diagnostic criteria Antiphospholipid syndrome: 2006 revision of the Sapporo APS classification criteria Acquired thrombotic thrombocytopenic purpura: consistent with a clinical diagnosis of TTP, including microscopic evidence of thrombocytopenia and red blood cell fragmentation (e.g., red blood cell fragmentation) 3. Multiple treatment regimens are ineffective or ineffective (including but not limited to high-dose glucocorticoids, adequate immunosuppressants and biologics) 4. Use of glucocorticoids (<=1mg/kg/d prednisone or equivalent doses of other hormones), DMARDs (such as methotrexate, hydroxychloroquine, azathioprine, mycophenolate mofetil, leflunomide, cyclosporine, etc.) must be on stable treatment for 4 weeks before receiving the first study drug, and no increase in hormone dose and other immunosuppressants throughout the study.

5. Subjects voluntarily participate in this study and voluntarily sign the informed consent form; 6. Subjects who have the possibility of having children or whose partners have the possibility of having children must agree to use effective contraception throughout the study period (but cannot use oral estrogen, use estrogen vaginal ring, etc.) 7. Additional enrollment criteria for different diseases (related to the degree of disease activity):

1. Patients with Behcet's disease must be active patients who meet the following conditions, and the active phase is defined as the emergence of new symptoms or the deterioration of existing symptoms, and one of the following conditions must be met:

   A. Organ involvement: involvement of any major organ (e.g., ocular lesions, vascular lesions, central nervous system, gastrointestinal system); B. 100% increase in the number of oral or genital ulcers >=compared to the onset of oral/genital ulcers compared to the first day; or an increase in the number of oral or genital ulcers by 3; C. Canker disease is at least 12 months; D. History of several oral ulcers per month E. Arthritis: >=50% increase in the number of swollen joints, or 3 more swollen joints; F. Skin lesions (non-oral/genital ulcers): >= physician overall lesion score increased by >=50% or by two points in the total score.
2. Patients with active inflammatory myopathy need to meet the following additional conditions:

   Active myositis as defined by the Baseline Freehand Muscle Strength Test (MMT-8) of no more than 125/150 and at least 2 additional CSMs that meet the criteria specified below:

   a) Visual Analogue Scale[VAS] of patient global activity ≥2 cm, b) physician's global disease activity ≥2 cm, c) Health Assessment Questionnaire (HAQ) Disability Index ≥ 0.25 d) Elevation of at least one muscle enzyme [including creatine kinase (CK), aldolase, lactate dehydrogenase (LDH), alanine aminotransferase (ALT), and aspartate aminotransferase (AST)] with a minimum level of 1.3 x upper limit of normal e) Global Extramuscular Disease Activity Score, with a minimum of 1.0 cm on a 10 cm VAS scale [This measure is a physician's comprehensive assessment based on the assessment of physique, skin, bone, gastrointestinal, lung, and cardiac activity scale activity scores using the Myositis Disease Activity Assessment Tool (MDAAT).

   f) To ensure that we are able to recruit patients with active DM with severe rash who may not meet the MMT-8 criteria above, we recommend the use of additional inclusion criteria so that the International Myositis Assessment and Clinical Study (IMACS) Improved Definition (DOI) can be achieved: 1) MDAAT > on the 10 cm VAS scale 3 cm skin VAS score, and 2) at least 3 of the above 5 criteria.
3. ANCA-associated vasculitis:

   A. Comply with GPA/MPA/EGPA classification standards; B. Patients with severe vasculitis activity (meeting at least one of the following conditions);

   a) Renal involvement is characterized by one of the following: i. Evidence of glomerulonephritis in any of the following situations: Renal biopsy shows focal necrotizing glomerulonephritis. Active urinary sediment characterized by glomerular hematuria and proteinuria ii. Patients with prior normal or no prior renal disease document, estimated glomerular filtration rate (eGFR) <50 ml/min/1.73 m2, and prior chronic kidney disease (eGFR <60 ml/min/1.73 m2) showed a reduction in eGFR of at least 25% compared with the previous one.

   b) Pulmonary hemorrhage due to active vasculitis satisfies all three of the following: i. Chest X-ray or CT scan showing diffuse pulmonary infiltrates ii. Pulmonary infiltrates that cannot be explained by other causes (e.g., volume overload or pulmonary infection) iii. At least one of the following: Evidence of alveolar hemorrhage on bronchoscopy or bloody bronchoalveolar lavage Hemoptysis was observed Unexplained anemia (<10 g/dL) or decreased hemoglobin (>1 g/dL) and less than 10g/dL Increased carbon dioxide dispersion
4. Additional Enrollment Criteria for Systemic Sclerosis:

   Subjects are at high risk of fatal outcomes based on the following prognostic factors: Subjects must have the following "a" , and at least one of "b" or "c".

   a) Diffuse cutaneous scleroderma with an mRSS score of >=16, validated by the same physician at 2 different times >= 1 day apart and separated by < 28 days.

   b) Presence of SSc-related lung disease with FVC < 70% or 70% predicted DLCO < after hemoglobin correction and evidence of alveolitis obtained by high-resolution chest CT scan or PAL.

   c) History of SSc-related nephropathy, no disease activity before enrollment screening. A history of hypertensive renal crisis with scleroderma is included in this criterion and is defined as follows: i. History of new-onset hypertension based on any of the following (must be repeated and confirmed at least 2 hours apart within 3 days of the first event) with change from baseline SBP>=140 mmHg DBP>=90 mmHg SBP rose by >=30 mmHg compared to baseline DBP increased by >=20 mmHg compared to baseline AND ii. One of the following 5 characteristics Serum creatinine increased >= >50% from baseline proteinuria: >=2+; Creatinine ratio > upper limit of normal Thrombocytopenia: <100, 000 plts/mm3 Hemolysis: increased by blood smear or reticulocyte count
5. Additional enrollment criteria for systemic lupus erythematosus A. The SLEDAI score of the patient before enrollment >= 7 points B. Failure to receive the following treatments: oral prednisone >=20 mg/d; Cyclophosphamide 0.4 to 0.6 g/m2 once every two weeks for 6 months, or other immunosuppressants such as mycophenolate mofetil 2 g/day for 3 months without remission.
6. Additional enrollment criteria for antiphospholipid syndrome A. Cardiolipin antibody, lupus anticoagulant factor, and anti-β2-glycoprotein 1 antibody were all positive before enrollment.

   B. History of thromboembolism or morbid pregnancy confirmed by clear objective evidence.
7. Sjögren's disease additional enrollment criteria A. Positive anti-Ro/SSA antibody screen. B. ESSDAI>= 6 POINTS
8. Additional enrollment criteria for IgG4-related diseases (confirmed: A+ B+C) A. Clinical examination showing the presence of characteristic diffuse/local swelling or masses in a single or multiple organs.

B. Blood tests show elevated serum IgG4 concentration (135 mg/dl). C. Histopathological examination shows significant lymphocytic and plasmacytic infiltration and fibrosis or IgG4+ plasmacyte infiltration (IgG4+/IgG+ cell ratio >40% and >10 IgG4+ plasma cells/HPF).

Exclusion Criteria:

1. Use of rituximab or other monoclonal antibodies within 1.6 months.
2. Received high-dose glucocorticoids (>1 mg/kg/d) within 1 month.
3. Serious complications: including heart failure (>= NYHA Class III), renal insufficiency (creatinine clearance <=30 ml/min), hepatic insufficiency (serum ALT or AST greater than three times the upper limit of normal, or total bilirubin greater than the upper limit of normal)
4. Other severe, progressive, or uncontrollable hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral diseases (including demyelinating diseases such as multiple sclerosis).
5. Known allergies, hyperreactivity, or intolerance to IL-2 or its excipients.
6. Have a serious infection (including but not limited to hepatitis, pneumonia, bacteremia, pyelonephritis, Epstein-Barr virus, tuberculosis infection), or hospitalization for infection, or use of intravenous antibiotics for treatment of infection 2 months prior to the first dose of treatment.
7. Chest imaging showing malignancy or current activity within 3 months prior to the first use of study drug Abnormalities in sexually transmitted infections (including tuberculosis).
8. Infection with HIV (HIV antibody-positive serology) or hepatitis C (Hep C antibody-positive serology).

If seropositive, it is advisable to consult a physician with expertise in the treatment of HIV or hepatitis C virus infection.

10. Any known malignancy or history of malignancy within the past 5 years (with the exception of non-melanoma skin cancer, non-melanoma skin cancer with no signs of recurrence or surgically cured cervical tumor within 3 months prior to the use of the first investigational agent).

11. Have an uncontrolled mental or emotional disorder, including a history of drug and alcohol abuse within the past 3 years, which may preclude the successful completion of the study.

12. Received or anticipated receipt of any live viral or bacterial vaccine injection within 3 months prior to the first injection of study dose, during the study, or within 4 months after the last injection of study dose. Bacillus Calmette-Guérin vaccination within 12 months of screening.

13. Pregnant, lactating women (WCBP) who are unwilling to use medically approved contraception during treatment and for 12 months after the end of treatment.

14. Males whose partner is of childbearing potential but who are unwilling to use appropriate medically approved contraception during treatment and for 12 months after the end of treatment.

15. Patients with inflammatory myopathies should additionally exclude: 3) Adolescent DM or PM, myositis overlaps with another connective tissue disease, cancer-associated myositis, inclusion body myositis, or any other non-immune-mediated myopathy.

4) Severe muscle impairment is defined as a baseline global muscle impairment score of MDI (Myositis Injury Index) >=5cm on 10 cm VAS.

16. ANCA-associated vasculitis requires additional exceptions: positive anti-GBM antibodies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Systemic Lupus Erythematosus primary outcome | From enrollment to the end of treatment at 24 weeks
  Percentage of SLE participants who had a response on the SLE Responder Index (SRI-4) at 24 weeks. The Systemic Lupus Erythematosus Responder Index-4 (SRI-4) was used to assess the treatment efficacy in systemic lupus erythematosus (SLE).The scale ranges from 0 to 105, with higher scores indicating worse disease activity. A response is defined as a ≥4-point improvement from baseline at 24 weeks
Sjogren syndrome primary outcome | From enrollment to the end of treatment at 24 weeks
  Proportion of participants with a Sjögren's Tool for Assessing Response (STAR) score of greater than or equal to five at 24 weeks. The STAR is a composite score used to evaluate the clinical response in patients with Sjögren's syndrome. The STAR score ranges from 0 to 9, with higher scores indicating better clinical response. A score of ≥5 at 24 weeks indicates a positive response to treatment.
Inflammatory Myopathy primary outcome | From enrollment to the end of treatment at 24 weeks
  TIS ranges from 0 to 100, with a higher score denoting greater improvement. In adults, TIS can be stratified into the following improvement categories for each patient at each timepoint (minimal improvement [TIS ≥20]; moderate improvement [TIS ≥40]; major improvement [TIS ≥60]). Thus, in the above example the patient would be classified as having moderate improvement [TIS ≥40].
Systemic Sclerosis primary outcome | From enrollment to the end of treatment at 24 weeks
  Change in the Modified Rodnan Skin Score (mRSS) at 24 weeks compared to baseline. The mRSS is a clinical tool used to assess the severity of skin thickening in patients with systemic sclerosis (scleroderma). The mRSS ranges from 0 to 51, with higher scores indicating more severe skin thickening. A decrease in the mRSS score indicates an improvement in skin involvement
Behçet's Disease primary outcome | From enrollment to the end of treatment at 24 weeks
  Proportion of participants with complete remission of oral ulcers at 24 weeks. Oral ulcer resolution is defined as the complete disappearance of all oral ulcers, as observed during clinical examination. A participant is considered to have achieved complete remission if no oral ulcers are present at the 24-week visit
ANCA associated Vasculitis primary outcome | From enrollment to the end of treatment at 52 weeks
  Proportion of participants achieving Birmingham Vasculitis Activity Score (BVAS) of 0 at 24 weeks. BVAS is a composite score used to assess disease activity in vasculitis, ranging from 0 to 63 or higher. Higher scores indicate more severe disease activity. A decrease in BVAS at 24 weeks indicates an improvement in disease activity.
Antiphospholipid Syndrome primary outcome | From enrollment to the end of treatment at 52 weeks
  Number and timing of thrombotic events occurring within 52 weeks.
Acquired Thrombotic Thrombocytopenic Purpura primary outcome | From enrollment to the end of treatment at 52 weeks
  Time to normalization of platelet count.
IgG4-related Disease primary outcome | From enrollment to the end of treatment at 24 weeks
  Proportion of participants with a decrease of greater than or equal to two points in the IgG4-related Disease Responder Index (IgG4RD RI) at 24 weeks compared to baseline. The IgG4RD RI is a composite score used to assess the response to treatment in IgG4-related disease. The score ranges from 0 to 63, with higher scores indicating worse disease activity. A decrease of ≥2 points at 24 weeks indicates a meaningful improvement in disease activity compared to baseline

SECONDARY OUTCOMES:
Systemic Lupus Erythematosus primary secondary Outcome | From enrollment to the end of treatment at 24 weeks
  Change in SLEDAI-2K at 24 weeks compared to baseline. The SLEDAI-2K is a composite index used to assess disease activity in systemic lupus erythematosus. The score ranges from 0 to 105, with higher scores indicating more severe disease activity. An improvement of ≥4 points in the SLEDAI-2K score at 24 weeks compared to baseline is considered a clinically meaningful response, reflecting a reduction in disease activity
Sjogren syndrome secondary outcome | From enrollment to the end of treatment at 24 weeks
  Change in the EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI) score at 24 weeks compared to baseline. The ESSDAI is a composite score used to assess disease activity in patients with Sjögren's syndrome. The score ranges from 0 to 123, with higher scores indicating more severe disease activity. A decrease in the ESSDAI score at 24 weeks compared to baseline indicates an improvement in disease activity.
Inflammatory Myopathy secondary outcome | From enrollment to the end of treatment at 24 weeks
  Change in the Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) score at 24 weeks compared to baseline. The CDASI is a composite score used to assess the severity and extent of skin involvement in patients with cutaneous dermatomyositis. The score ranges from 0 to 132, with higher scores indicating more severe disease activity. A decrease in the CDASI score at 24 weeks compared to baseline indicates an improvement in skin involvement and disease severity.
Systemic Sclerosis secondary outcome | From enrollment to the end of treatment at 24 weeks
  Change in the Health Assessment Questionnaire Disability Index (HAQDI) score at 24 weeks compared to baseline. The HAQDI is a widely used measure of disability in patients with chronic diseases, assessing the impact of disease on daily functioning. The score ranges from 0 to 3, with higher scores indicating greater disability and more severe functional impairment. A decrease in the HAQDI score at 24 weeks compared to baseline indicates an improvement in the patient's functional status and a reduction in disability.
Behçet's Disease secondary outcome | From enrollment to the end of treatment at 24 weeks
  Change in the Behçet's Syndrome Activity Score (BSAS) at 24 weeks compared to baseline. The BSAS is a composite score used to assess the disease activity in patients with Behçet's syndrome, considering both clinical signs and symptoms. The score ranges from 0 to 85, with higher scores indicating greater disease activity and more severe symptoms. A decrease in the BSAS at 24 weeks compared to baseline indicates a reduction in disease activity and an improvement in clinical symptoms.
ANCA associated Vasculitis secondary outcome | From enrollment to the end of treatment at 52 weeks
  Change in the Birmingham Vasculitis Activity Score (BVAS) at 52 weeks compared to baseline. The BVAS is a composite score used to assess the disease activity in patients with vasculitis. The score ranges from 0 to 63, with higher scores indicating greater disease activity. A decrease in the BVAS at 52 weeks compared to baseline indicates a reduction in disease activity and an improvement in clinical symptoms.
Antiphospholipid Syndrome secondary outcome | From enrollment to the end of treatment at 52 weeks
  Number and timing of bleeding events occurring within 52 weeks.
Acquired Thrombotic Thrombocytopenic Purpura secondary outcome | From enrollment to the end of treatment at 52 weeks
  Time to relapse of thrombotic thrombocytopenic purpura (TTP) within 52 weeks.
IgG4-related Disease secondary outcome | From enrollment to the end of treatment at 24 weeks
  IgG4-related Disease Responder Index (IgG4RD RI) scores at each follow-up visit. The IgG4RD RI is a composite index used to assess the response to treatment in patients with IgG4-related disease (IgG4-RD). The score is based on the evaluation of clinical symptoms, laboratory markers, and imaging results. The IgG4RD RI score ranges from 0 to 63, with higher scores indicating greater disease activity and worse outcomes. A decrease in the IgG4RD RI score at follow-up visits compared to baseline suggests improvement in disease activity and response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Peking University Institute of Rheuamotology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China